CLINICAL TRIAL: NCT06560151
Title: Randomized, Double-Blind, Phase 2 Study to Assess Safety and Immunogenicity of A/H5 Inactivated Monovalent Influenza Vaccines at Different Antigen Dose Levels Adjuvanted With AS03® or MF59®
Brief Title: Assess Safety and Immunogenicity of A/H5 Inactivated Monovalent Influenza Vaccines at Different Antigen Dose Levels Adjuvanted With AS03 or MF59
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Biomedical Advanced Research and Development Authority (U.S. Federal Agency)
Collaborators: Rho Federal Systems Division, Inc. (Industry); ICON plc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: BP-I-23-001
Record Dates: First submitted 2024-08-15; First posted 2024-08-19 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-12

CONDITIONS: Influenza
Keywords: A/H5; H5; Inactivated; Monovalent; Influenza; Vaccines; AS03; MF59
MeSH Terms: conditions — Influenza, Human | interventions — MF59 oil emulsion

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (15):
- Treatment Group A (Experimental): This treatment group of 60 participants (ages 18-64) in Treatment Group A will receive 3.75 µg of Egg-A/Astrakhan/3212/2020 (H5N8) antigen adjuvanted with a full dose of AS03A.
  Interventions: Biological: 3.75 µg H5N8 antigen plus full dose AS03A
- Treatment Group B (Experimental): This treatment group of 120 participants (60 participants ages 18-64 and 60 participants ages ≥65) in Treatment Group B will receive 7.5 µg of Egg-A/Astrakhan/3212/2020 (H5N8) adjuvanted with a full dose of AS03A.
  Interventions: Biological: 7.5 µg H5N8 antigen plus full dose AS03A
- Treatment Group C (Experimental): This treatment group of 120 participants (60 participants ages 18-64 and 60 participants age ≥65) will receive 15 µg of Egg-A/Astrakhan/3212/2020 (H5N8) adjuvanted with a full dose of AS03A.
  Interventions: Biological: 15 µg H5N8 antigen plus full dose AS03A
- Treatment Group D (Experimental): This treatment group of 60 participants (ages 18-64) will receive 3.75 µg of Egg-A/Astrakhan/3212/2020 (H5N8) adjuvanted with a half dose of AS03A.
  Interventions: Biological: 3.75 µg H5N8 antigen plus half dose AS03A
- Treatment Group E (Experimental): This treatment group of 120 participants (60 participants ages 18-64 and 60 participants age ≥65) will receive 7.5 µg of Egg-A/Astrakhan/3212/2020 (H5N8) adjuvanted with a half dose of AS03A.
  Interventions: Biological: 7.5 µg H5N8 antigen plus half dose AS03A
- Treatment Group F (Experimental): This treatment group of 120 participants (60 participants ages 18-64 and 60 participants age ≥65 will receive 15 µg of Egg-A/Astrakhan/3212/2020 (H5N8) adjuvanted with a half dose of AS03A.
  Interventions: Biological: 15 µg H5N8 antigen plus half dose AS03A
- Treatment Group G (Experimental): This treatment group of 60 participants (ages 18-64) will receive 3.75 µg of Egg-A/Astrakhan/3212/2020 (H5N8) adjuvanted with MF59.
  Interventions: Biological: 3.75 µg H5N8 antigen plus MF59
- Treatment Group H (Experimental): This treatment group of 120 participants (60 participants ages 18-64 and 60 participants age ≥65) will receive 7.5 µg of Egg-A/Astrakhan/3212/2020 (H5N8) adjuvanted with MF59.
  Interventions: Biological: 7.5 µg H5N8 antigen plus MF59
- Treatment Group I (Experimental): This treatment group of 120 participants (60 participants ages 18-64 and 60 participants age ≥65) will receive 15 µg of Egg-A/Astrakhan/3212/2020 (H5N8) adjuvanted with MF59.
  Interventions: Biological: 15 µg H5N8 antigen plus MF59
- Treatment Group J (Experimental): This treatment group of 60 participants (ages 18-64) will receive 3.75 µg of Egg-A/bar-headed goose/Qinghai Lake/1A/2005 (H5N1) adjuvanted with a full dose of AS03A.
  Interventions: Biological: 3.75 µg H5N1 antigen plus full dose AS03A
- Treatment Group K (Experimental): This treatment group of 120 participants (60 participants ages 18-64 and 60 participants age ≥65) will receive 7.5 µg of Egg-A/bar-headed goose/Qinghai Lake/1A/2005 (H5N1) adjuvanted with a full dose of AS03A.
  Interventions: Biological: 7.5 µg H5N1 antigen plus full dose AS03A
- Treatment Group L (Experimental): This treatment group of 60 participants (ages ≥65) will receive 15 µg of Egg-A/bar-headed goose/Qinghai Lake/1A/2005 (H5N1) adjuvanted with a full dose of AS03A.
  Interventions: Biological: 15 µg H5N1 antigen plus full dose AS03A
- Treatment Group M (Experimental): This treatment group of 60 participants (ages 18-64) will receive 3.75 µg of Egg-A/bar-headed goose/Qinghai Lake/1A/2005 (H5N1) adjuvanted with MF59.
  Interventions: Biological: 3.75 µg H5N1 antigen plus MF59
- Treatment Group N (Experimental): This treatment group of 120 participants (60 participants ages 18-64 and 60 participants age ≥65) will receive 7.5 µg of Egg-A/bar-headed goose/Qinghai Lake/1A/2005 (H5N1) adjuvanted with MF59.
  Interventions: Biological: 7.5 µg H5N1 antigen plus MF59
- Treatment Group O (Experimental): This treatment group of 60 participants (age ≥65) will receive 15 µg of Egg-A/bar-headed goose/Qinghai Lake/1A/2005 (H5N1) adjuvanted with MF59.
  Interventions: Biological: 15 µg H5N1 antigen plus MF59

INTERVENTIONS:
Biological: 3.75 µg H5N8 antigen plus full dose AS03A — Two intramuscular doses (21 days apart) of AS03A adjuvanted H5N8 vaccine.
  Arms: Treatment Group A
Biological: 7.5 µg H5N8 antigen plus full dose AS03A — Two intramuscular doses (21 days apart) of AS03A adjuvanted H5N8 vaccine.
  Arms: Treatment Group B
Biological: 15 µg H5N8 antigen plus full dose AS03A — Two intramuscular doses (21 days apart) of AS03A adjuvanted H5N8 vaccine.
  Arms: Treatment Group C
Biological: 3.75 µg H5N8 antigen plus half dose AS03A — Two intramuscular doses (21 days apart) of AS03A adjuvanted H5N8 vaccine.
  Arms: Treatment Group D
Biological: 7.5 µg H5N8 antigen plus half dose AS03A — Two intramuscular doses (21 days apart) of AS03A adjuvanted H5N8 vaccine.
  Arms: Treatment Group E
Biological: 15 µg H5N8 antigen plus half dose AS03A — Two intramuscular doses (21 days apart) of AS03A adjuvanted H5N8 vaccine.
  Arms: Treatment Group F
Biological: 3.75 µg H5N8 antigen plus MF59 — Two intramuscular doses (21 days apart) of MF59 adjuvanted H5N8 vaccine.
  Arms: Treatment Group G
Biological: 7.5 µg H5N8 antigen plus MF59 — Two intramuscular doses (21 days apart) of MF59 adjuvanted H5N8 vaccine.
  Arms: Treatment Group H
Biological: 15 µg H5N8 antigen plus MF59 — Two intramuscular doses (21 days apart) of MF59 adjuvanted H5N8 vaccine.
  Arms: Treatment Group I
Biological: 3.75 µg H5N1 antigen plus full dose AS03A — Two intramuscular doses (21 days apart) of AS03A adjuvanted H5N1 vaccine.
  Arms: Treatment Group J
Biological: 7.5 µg H5N1 antigen plus full dose AS03A — Two intramuscular doses (21 days apart) of AS03A adjuvanted H5N1 vaccine.
  Arms: Treatment Group K
Biological: 15 µg H5N1 antigen plus full dose AS03A — Two intramuscular doses (21 days apart) of AS03A adjuvanted H5N1 vaccine.
  Arms: Treatment Group L
Biological: 3.75 µg H5N1 antigen plus MF59 — Two intramuscular doses (21 days apart) of MF59 adjuvanted H5N1 vaccine.
  Arms: Treatment Group M
Biological: 7.5 µg H5N1 antigen plus MF59 — Two intramuscular doses (21 days apart) of MF59 adjuvanted H5N1 vaccine.
  Arms: Treatment Group N
Biological: 15 µg H5N1 antigen plus MF59 — Two intramuscular doses (21 days apart) of MF59 adjuvanted H5N1 vaccine.
  Arms: Treatment Group O

SUMMARY:
This BARDA-sponsored, randomized, double-blind, phase 2 study is designed to assess safety and immunogenicity of A/H5 inactivated monovalent influenza vaccines at different antigen dose levels adjuvanted with AS03 or MF59.

DETAILED DESCRIPTION:
This is a randomized, double-blind, phase 2 study to assess safety and immunogenicity of egg-based H5N8 and H5N1 influenza vaccines at different antigen dose levels (3.75, 7.5, and 15 μg) adjuvanted with AS03A full dose, AS03A half dose (H5N8 only), or MF59. AS03A is the adjuvant AS03®. Healthy adult male and female (non-pregnant) participants, aged 18 years and older, will be screened for baseline health status to ensure trial eligibility. Participants meeting all the inclusion and none of the exclusion criteria will be randomized to receive vaccine doses according to treatment groups defined by antigen (H5N1 or H5N8), antigen dose level (3.75, 7.5, and 15 μg), and adjuvant (AS03A full dose, AS03A half dose, or MF59). Two doses of adjuvanted vaccine separated by 21 days will be administered to approximately 1380 participants, including 780 participants 18 through 64 years old who will be randomized equally to 1 of 13 treatment groups (A, B, C, D, E, F, G, H, I, J, K, M, and N), and 600 participants ≥65 years old who will be randomized equally to 1 of 10 treatment groups (B, C, E, F, H, I, K, L, N, and O).

Safety assessments will be based on solicited Adverse Events (AEs) (local and systemic reactogenicity symptoms) with onset within 8 days following each vaccination, inclusive of the vaccination day (Day 1 through Day 8 and Day 22 through Day 29); unsolicited Treatment Emergent Adverse Events (TEAEs) with onset within 22 days following each vaccination, inclusive of the vaccination day (Day 1 through Day 22 and Day 22 through Day 43); and treatment-emergent Serious Adverse Events (SAEs), Potential Immune-Mediated Diseases (pIMDs), and Medically Attended Adverse Events (MAAEs) occurring during study participation (through Day 203). Immunogenicity assessments will include titer, seroprotection rate, and seroconversion rate based on serum Hemagglutination Inhibition (HAI) antibodies, and titer and seroconversion rate based on serum microneutralization (MN) antibodies. Study vaccines will be prepared and administered by unblinded personnel. All other trial assessments will be performed only by blinded personnel.

ELIGIBILITY:
Inclusion Criteria:

1. Male or non-pregnant female, 18 years of age or older at the time of screening and informed consent.
2. Willing and able to provide written informed consent prior to initiation of study procedures.
3. Agrees to have specimens collected during this trial specifically for the purpose of future research stored for future research use.
4. In relatively stable health, as determined by medical history and physical examination.

   a. Any chronic medical diagnoses or conditions should be stable and well managed, with no significant changes expected during the study period, and in the opinion of the site investigator, will not impact the ability to assess safety and/or immunogenicity per the study design.
5. If a female of childbearing potential who is sexually active, agrees to use an adequate method of birth control from Screening through 4 weeks following the last study vaccination and has used an adequate birth control method for at least 2 months prior to Screening.

   a. Female of childbearing potential is defined as post onset menarche and pre-menopausal person capable of becoming pregnant. This does not include females who meet any of the following conditions:

   i. menopausal >2 years

   ii. tubal ligation >1 year

   iii. bilateral salpingo-oophorectomy

   iv. hysterectomy.

   b. Adequate contraception is defined as a contraceptive method with a failure rate of less than 1% per year when used consistently and correctly and when applicable, in accordance with the product label, for example: oral contraceptives, either combined or progestogen alone; injectable progestogen; implants of etonogestrel or levonorgestrel; estrogenic vaginal ring; percutaneous contraceptive patches; intrauterine device or intrauterine system; the female participant has exclusively female sexual partners; male partner is sterile or otherwise unable to produce sperm (information on the person's sterility can come from the site personnel's review of the participant's medical records or interview with the participant regarding her medical history); male condom combined with a vaginal spermicide (foam, gel, film, cream, or suppository); or male condom combined with a female diaphragm, either with or without a vaginal spermicide (foam, gel, film, cream, or suppository).
6. Available for all study visits, willing to participate in all study procedures, and not planning to relocate from the area for the duration of the study.

Exclusion Criteria:

1. Has an acute illness, as determined by the site investigator, within 72 hours prior to vaccination.

   a. An acute illness that is nearly resolved, with only minor residual symptoms remaining, is allowable if, in the opinion of the site investigator, the residual symptoms will not interfere with the ability of study staff to assess safety parameters as required by the protocol.
2. Has a history of severe reaction to any influenza vaccine.
3. Has a known allergy to squalene-based adjuvants.
4. Female of childbearing potential who has a positive urine pregnancy test or who is currently breastfeeding.
5. Has a body mass index >35 kg/m2 .
6. Has known human immunodeficiency virus, hepatitis B, or hepatitis C infection (based on medical history).
7. Has a history of any pIMDs (list provided in Protocol Appendix 3), neuralgia, paresthesia, neuritis, convulsions, or encephalomyelitis within 90 days prior to Screening, or a family history of Guillain-Barré syndrome.
8. Has narcolepsy or a first degree relative with narcolepsy.
9. Has a history of alcohol or drug abuse within 5 years prior to Screening.
10. Has any diagnosis, current or past, of schizophrenia, bipolar disease, or any other psychiatric diagnosis that may, in the opinion of the site investigator, interfere with participant compliance or safety evaluations.
11. Is immunosuppressed due to an underlying disease or medication, use of anticancer chemotherapy (cytotoxic), or radiation therapy.
12. With the exception of basal or squamous cell skin cancer, has known active neoplastic disease, including hematologic malignancy.
13. Has long-term use (≥14 consecutive days) of glucocorticoids including oral or parenteral prednisone or prednisone equivalent (>20 mg total dose per day) or high-dose inhaled steroids (>800 µg/day of beclomethasone dipropionate or equivalent) within 1 month prior to screening in this study. However, participants on low-dose inhaled steroids (≤800 µg/day of beclomethasone dipropionate or equivalent) or topical steroids are not excluded.
14. Has received immunoglobulin or other blood product (with the exception of Rho[D] immune globulin) within the 90 days prior to screening in this study.
15. Has received any (licensed or under Emergency Use Authorization [EUA]) live vaccines within 4 weeks or inactivated, messenger RNA (mRNA), or recombinant protein vaccines within 2 weeks prior to screening, or plans to receive such vaccines (including seasonal influenza and COVID-19 vaccines) from screening through 22 days following the second dose of the study vaccine, inclusive of the vaccination day (Screening Visit through Day 43).
16. Is participating or plans to participate in another interventional clinical trial (either active or follow-up phase) during the study period.
17. Has participated in an A(H5) influenza vaccine study in the past or has a history of A(H5) influenza infection prior to vaccination in this study. This includes, but is not limited to, influenza sub-types A(H5N1), A(H5N8), and A(H5N6).
18. Has any laboratory test result or clinical findings (including vital signs) that singly or in combination are likely to unfavorably alter the risks of participant participation or to confound study safety or immunogenicity results, in the opinion of the site investigator. Additionally, the following are exclusionary:

    1. Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >2 times the upper limit of normal (ULN), or
    2. Bilirubin >1.5 times the ULN unless isolated Gilbert's syndrome.
19. Has any disease or medical condition that, in the opinion of the site investigator, might confound interpretation of safety or immunogenicity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1380 (Actual)
Dates: Start 2024-08-21 (Actual); Primary Completion 2025-01-02 (Actual); Study Completion 2025-06-11 (Actual)

PRIMARY OUTCOMES:
The percentage of participants who experience any solicited local reactogenicity symptom occurring within 8 days of each vaccination, inclusive of the vaccination day. | Day 1 through Day 8 and Day 22 through Day 29
The percentage of participants who experience any solicited systemic reactogenicity symptom occurring within 8 days of each vaccination, inclusive of the vaccination day. | Day 1 through Day 8 and Day 22 through Day 29
The percentage of participants achieving seroprotection at Day 43 based on serum HAI antibody titers (≥1:40) to A/Astrakhan (H5N8). | Day 43

SECONDARY OUTCOMES:
The percentage of participants who experience any unsolicited TEAE within 22 days of each vaccination, inclusive of the vaccination day. | Day 1 through Day 22 and Day 22 through Day 43
The percentage of participants who experience any treatment-emergent SAE. | Day 1 through Day 203
The percentage of participants who experience any treatment-emergent MAAE. | Day 1 through Day 203
The percentage of participants who experience any treatment-emergent pIMD. | Day 1 through Day 203
The percentage of participants achieving seroprotection at Day 43 based on serum HAI antibody titers (≥1:40) to A/bar-headed goose (H5N1). | Day 43
Serum HAI antibody titers to A/Astrakhan (H5N8) at Screening. | Screening
Serum HAI antibody titers to A/Astrakhan (H5N8) at Day 22. | Day 22
Serum HAI antibody titers to A/Astrakhan (H5N8) at Day 43. | Day 43
Serum HAI antibody titers to A/Astrakhan (H5N8) at Day 203. | Day 203
Serum HAI antibody titers to A/bar-headed goose (H5N1) at Screening. | Screening
Serum HAI antibody titers to A/bar-headed goose (H5N1) at Day 22. | Day 22
Serum HAI antibody titers to A/bar-headed goose (H5N1) at Day 43. | Day 43
Serum HAI antibody titers to A/bar-headed goose (H5N1) at Day 203 | Day 203
The percentage of participants achieving seroprotection at Day 22 based on serum HAI antibody titers (≥1:40) to A/Astrakhan (H5N8). | Day 22
The percentage of participants achieving seroprotection at Day 203 based on serum HAI antibody titers (≥1:40) to A/Astrakhan (H5N8). | Day 203
The percentage of participants achieving seroprotection at Day 22 based on serum HAI antibody titers (≥1:40) to A/bar-headed goose (H5N1). | Day 22
The percentage of participants achieving seroprotection at Day 203 based on serum HAI antibody titers (≥1:40) to A/bar-headed goose (H5N1). | Day 203
The percentage of participants achieving seroconversion at Day 22 based on serum HAI antibody titers to A/Astrakhan (H5N8). | Day 22
The percentage of participants achieving seroconversion at Day 43 based on serum HAI antibody titers to A/Astrakhan (H5N8). | Day 43
The percentage of participants achieving seroconversion at Day 203 based on serum HAI antibody titers to A/Astrakhan (H5N8). | Day 203
The percentage of participants achieving seroconversion at Day 22 based on serum HAI antibody titers to A/bar-headed goose (H5N1). | Day 22
The percentage of participants achieving seroconversion at Day 43 based on serum HAI antibody titers to A/bar-headed goose (H5N1). | Day 43
The percentage of participants achieving seroconversion at Day 203 based on serum HAI antibody titers to A/bar-headed goose (H5N1). | Day 203
Serum MN antibody titers to A/Astrakhan (H5N8) at Screening. | Screening
Serum MN antibody titers to A/Astrakhan (H5N8) at Day 22. | Day 22
Serum MN antibody titers to A/Astrakhan (H5N8) at Day 43. | Day 43
Serum MN antibody titers to A/Astrakhan (H5N8) at Day 203. | Day 203
Serum MN antibody titers to A/bar-headed goose (H5N1) at Screening. | Screening
Serum MN antibody titers to A/bar-headed goose (H5N1) at Day 22. | Day 22
Serum MN antibody titers to A/bar-headed goose (H5N1) at Day 43. | Day 43
Serum MN antibody titers to A/bar-headed goose (H5N1) at Day 203. | Day 203
The percentage of participants achieving seroconversion at Day 22 based on serum MN antibody titers to A/Astrakhan (H5N8). | Day 22
The percentage of participants achieving seroconversion at Day 43 based on serum MN antibody titers to A/Astrakhan (H5N8). | Day 43
The percentage of participants achieving seroconversion at Day 203 based on serum MN antibody titers to A/Astrakhan (H5N8). | Day 203
The percentage of participants achieving seroconversion at Day 22 based on serum MN antibody titers to A/bar-headed goose (H5N1). | Day 22
The percentage of participants achieving seroconversion at Day 43 based on serum MN antibody titers to A/bar-headed goose (H5N1). | Day 43
The percentage of participants achieving seroconversion at Day 203 based on serum MN antibody titers to A/bar-headed goose (H5N1). | Day 203

CONTACTS AND LOCATIONS:
Locations (20):
- United States (20):
  - DelRicht Research - Atlanta, Atlanta, Georgia
  - Javara Research - Privia Medical Group Georgia, Savannah, Georgia
  - Accellacare - Duly Health and Care - Oak Lawn, Oak Lawn, Illinois
  - Johnson County Clin-Trials (JCCT), Lenexa, Kansas
  - Alliance for Multispecialty Research - Wichita East - Heartland Research Associates, Wichita, Kansas
  - Alliance for Multispecialty Research - Lexington, Lexington, Kentucky
  - DelRicht Research - New Orleans - Prytania Street, New Orleans, Louisiana
  - DelRicht Research - Prairieville, Prairieville, Louisiana
  - Rochester Clinical Research, New York, New York
  - Accellacare - Cary, Cary, North Carolina
  - Accellacare of Hickory, Hickory, North Carolina
  - Accellacare - Piedmont Healthcare, Statesville, North Carolina
  - Accellacare - Tradd Court, Wilmington, North Carolina
  - CTI Clinical Research Center, Cincinnati, Ohio
  - DelRicht Research - Tulsa, Tulsa, Oklahoma
  - Tekton Research - Oklahoma - Primary Health Partners, Yukon, Oklahoma
  - Tekton Research - Austin, Austin, Texas
  - Javara Research - Privia Medical Group Gulf Coast, Conroe, Texas
  - Tekton Research - San Antonio, San Antonio, Texas
  - DelRicht Research - Virgina, Sterling, Virginia

DOCUMENTS (1):
  • Informed Consent Form (2024-08-19): https://cdn.clinicaltrials.gov/large-docs/51/NCT06560151/ICF_000.pdf